CLINICAL TRIAL: NCT04882007
Title: Randomized, Double-blind, Phase 2 Study to Evaluate the Efficacy and the Safety of OSE-127 Versus Placebo in Subjects With Moderate to Severe Active Ulcerative Colitis Who Have Failed or Are Intolerant to Previous Treatment(s)
Brief Title: Study of OSE-127 vs Placebo in Patients With Moderate to Severe Active Ulcerative Colitis
Acronym: CoTikiS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OSE Immunotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OSE-127-C201; 2020-001398-59 (EudraCT Number)
Record Dates: First submitted 2021-04-13; First posted 2021-05-11 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-03

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis; inflammatory bowel diseases; Auto-Immune Diseases; CD127/IL-7Rα Antagonist
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During the Double-blind phase all participants will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- OSE-127 High dose induction phase (Experimental): OSE-127 mAb antagonist to CD127 receptor (or IL-7Rα) intravenous infusion 3 total infusions, weeks 0, 2, and 6
  Interventions: Drug: OSE-127
- OSE-127 Low dose induction phase (Experimental): OSE-127 mAb antagonist to CD127 receptor (or IL-7Rα) intravenous infusion 3 total infusions, weeks 0, 2, and 6
  Interventions: Drug: OSE-127
- Placebo induction phase (Placebo Comparator): Normal saline intravenous infusion 3 total infusions, weeks 0, 2, and 6
  Interventions: Drug: Placebo
- OSE-127 High dose optional extension phase (Experimental): OSE-127 mAb antagonist to CD127 receptor (or IL-7Rα) intravenous infusion 7 total infusions, weeks 10, 14, 18, 22, 26, 30, and 34
  Interventions: Drug: OSE-127

INTERVENTIONS:
Drug: OSE-127 — mAb antagonist to CD127 receptor (or IL-7Rα)
  Arms: OSE-127 High dose induction phase; OSE-127 High dose optional extension phase; OSE-127 Low dose induction phase
Drug: Placebo — Normal saline
  Arms: Placebo induction phase

SUMMARY:
This is a phase 2, multicenter, randomized, double-blind, placebo-controlled, parallel-group study in patients with moderate to severe active ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent document indicating that the patient has been informed of all the pertinent aspects of the trial prior to enrollment
2. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
3. Willingness to refrain from live or attenuated vaccines during the study and for 12 weeks after last dose
4. Male or female 18 to 75 years of age, inclusive
5. Diagnosis of moderate to severe active UC made at least 3 months before the screening visit. The diagnosis of UC must have been confirmed by endoscopy, with a minimal extent of 15 cm from anal margin and histology (Moderate to severe active UC is defined by a modified Mayo score between 4 and 9, inclusive. The modified Mayo score is defined by the addition of the rectal bleeding subscore, the stool frequency sub-score, and the endoscopic sub-score. Thus, to be included, a patient must have the following:

   1. a rectal bleeding score ≥ 1,
   2. a stool frequency score ≥ 1 (sub-score calculated before bowel preparation), and
   3. an endoscopic sub-score ≥ 2
6. No previous biologic therapy (i.e., TNF antagonists, vedolizumab or ustekinumab) and prior or current UC documented medication history that includes at least 1 of the following:

   1. Corticosteroids
   2. Immunosuppressive agents

OR

Previous or current biologic therapy

Exclusion Criteria:

1. Stoma, proctocolectomy, or subtotal colectomy
2. Physician judgment that patient is likely to require any surgery for UC during the study duration, or double-blind phase duration at least
3. Evidence of fulminant colitis, toxic megacolon, or perforation
4. Current or recent (within 4 weeks prior to screening) hospitalization for UC care and/or treatment with IV steroids
5. The following laboratory results at screening:

   1. Elevation at screening of aminotransferase (AST), alanine aminotransferase (ALT) > 3 × the upper limit of normal (ULN) or total bilirubin > 2 × ULN (unless due to Gilbert's disease) or evidence of chronic liver disease
   2. Platelet count < 100,000/mm3
   3. Hemoglobin (Hgb) < 8.5 g/dL
   4. Neutrophils < 1500/mm3
   5. Lymphocytes < 800/mm3
   6. Absolute white blood cell (WBC) count < 3000/mm3
6. Crohn's disease or indeterminate colitis or any other diagnosis not consisting with UC
7. History or evidence of incompletely resected colonic dysplasia or unconventional lesion at risk of colonic adenocarcinoma
8. Stool culture or other examination positive for enteric pathogen, including Clostridium difficile (C. diff) toxin. If positive, the patient should be treated and rescreening is allowed.
9. Men or women with childbearing potential not willing to use adequate birth control during the study. Adequate birth control includes surgical sterilization, intrauterine device, oral contraceptive, contraceptive patch, long-acting injectable contraceptive, partner's vasectomy, double-barrier method (condom, diaphragm with spermicide), or abstinence during study and 30 days following the last follow-up visit. Women of childbearing potential will enter the study after a negative pregnancy test.
10. Breastfeeding
11. Chronic use of nonsteroidal anti-inflammatory drugs (NSAIDs) from screening through the end of the study
12. Use of topical steroids and/or topical 5-aminosalicylic acid preparations within 2 weeks before the screening visit (all such medications should be withdrawn at least 2 weeks prior to the screening visit)
13. Use of antidiarrheals within 2 weeks before the screening visit (all such medications should be withdrawn at least 2 weeks prior to the screening visit)
14. Treatment with azathioprine, 6-MP, methotrexate (MTX), cyclosporin, tacrolimus, sirolimus, leflunomide and/or mycophenolate mofetil within 4 weeks before the screening visit (all such medications should be withdrawn at least 4 weeks prior to the screening visit)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Change in modified Mayo Score | Baseline and Week 10
  Change in modified Mayo Score between baseline and Week 10 clinical symptoms (stool frequency and rectal bleeding sub-scores) additionally to the endoscopic sub-score

SECONDARY OUTCOMES:
Clinical Remission | Week 10
  Number and proportion of patients achieving clinical remission at Week 10, defined as a modified Mayo score of ≤ 2 points and with no individual sub-score of > 1 point and a rectal bleeding at 0, therefore a stool frequency score of 0 or 1 and an endoscopic score of 0 or 1
Clinical efficacy of OSE-127 vs placebo | Week 10
  Number and proportion of patients with a clinical response defined as a reduction in the modified Mayo score of ≥ 3 points and of ≥ 30% from baseline, with an accompanying decrease from baseline in the rectal bleeding sub-score of ≥ 1 point or an absolute rectal bleeding sub-score of ≤ 1 point
Efficacy of OSE-127 vs placebo on endoscopic remission | Week 10
  Number and proportion of patients with an endoscopic remission defined by an endoscopic Mayo sub-score =0
Efficacy of OSE-127 vs placebo on endoscopic improvement | Week 10
  Number and proportion of patients with endoscopic response or improvement defined by an endoscopic subscore of Mayo ≤ 1 point
Efficacy of OSE-127 vs placebo on endoscopic improvement | Week 10
  Mean change from baseline in the endoscopic activity measured by the Ulcerative Colitis Endoscopic Index of Severity (UCEIS)
Overall safety and tolerability of OSE-127 in patients with moderate to severe UC | Week 0 to Week 22 for patients not participating in the optional extension, and Week 0 to Week 50 for patients participating in the optional extension
  Frequency and severity of reported treatment-emergent adverse events, serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Comis, MD, Study Director — OSE Immunotherapeutics
Locations (55):
- Belarus (5):
  - Brest Regional Hospital, Brest
  - Grodno University Hospital, Grodno
  - Gomel Regional Clinical Hospital, Homyel
  - City Clinical Emergency Hospital, Minsk
  - Vitebsk Regional Clinical Hospital, Vitebsk
- Belgium (3):
  - UZ Leuven - Department of Gastroenterology and Hepatology, Leuven
  - CHU Liège, Liège
  - Groupe Santé CHC - Clinique du Mont Légia, Liège
- Bulgaria (10):
  - Medical Center Medconsult Pleven - OOD, Pleven
  - Medical Center Medconsult Pleven, Pleven
  - Acibadem City Clinic University Multiprofile Hospital for Active Treatment - EOOD, Clinic of Gastroenterology, Sofia
  - Medical Center Asklepion - Researches in humane medicine (EOOD), Sofia
  - Medical Center Asklepion, Sofia
  - Medical Center Hera EOOD, Sofia
  - Medical Center Hera, Sofia
  - UMHAT Tsaritsa Yoanna - ISUL - EAD, Sofia
  - Medical center VIP Clinic - OOD, Varna
  - Medical Center VIP Clinic, Varna
- University Hospital Center Split, Split, Croatia
- Georgia (6):
  - EVEX Hospitals JSC, Kutaisi
  - West Regional Center of Modern Medical Technologies Ltd, Kutaisi
  - Institute of Clinical Cardiology, Tbilisi
  - Israel-Georgia Medical Research Clinic Helsicore Ltd, Tbilisi
  - JSC Clinic Jerarsi, Tbilisi
  - Multiprofile Clinic Consilium Medulla Ltd, Tbilisi
- Hungary (3):
  - Clinexpert SMO, Budapest
  - II. Sz. Belgyogyaszati Klinika, Semmelweis Egyetem, Budapest
  - II. Sz Belgyogyasztai Intezet, Gasztroenterologia Debreceni Egyetem, Debrecen
- Latvia (4):
  - Polana-D, Daugavpils
  - Liepāja Regional Hospital, Liepāja
  - Digestive Diseases Centre GASTRO, Riga
  - Pauls Stradins Clinical University Hospital, Riga
- Poland (7):
  - Centrum Opieki Zdrowotnej Orkan-med, Ksawerów
  - Centrum Medyczne Med-Gastr, Lodz
  - Oddział Kliniczny Gastroenterologii Ogólnej i Onkologicznej, Lodz
  - Medicome Sp. z o.o., Oświęcim
  - Centrum Medyczne Medyk, Rzeszów
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Melita Medical, Wroclaw
- Russia (7):
  - Prof. S.V. Ochapovskiy Regional Clinical Hospital No.1, Krasnodar
  - Ryzhikh State Coloproctology Research Center, Moscow
  - LLC Novosibirskiy Gastrocenter, Novosibirsk
  - Medical Center Healthy Family LLC, Novosibirsk
  - State Budgetary Healthcare Institution of the Stavropol Region - Pyatigorsk Oncology Dispensary, Pyatigorsk
  - Saratov State Medical University, Saratov
  - Ekaterinburg City Clinical Hospital No. 14, Yekaterinburg
- 301 Fairfield Medical Suite, Cape Town, South Africa
- Ukraine (8):
  - Dnipropetrovsk I.I. Mechnikov Regional Clinical Hospital - Dnipropetrovsk Regional Council, Dnipro
  - Prof. O.O. Salimov City Clinical Hospital #2 - Kharkiv City Council, Kharkiv
  - Kryvyi Rih City Clinical Hospital #2, Kryvyi Rih
  - Kyiv Regional Clinical Hospital - Kyiv Regional Council, Kyiv
  - Medical Center OK!Clinic+ of International Institute of Clinical Studies LLC, Kyiv
  - Ternopil University Hospital - Ternopil Regional Council, Ternopil
  - Andrii Novak Transcarpathian Regional Clinical Hospital, Uzhhorod
  - Municipal Institution City Clinical Hospital #6 - Therapeutic Department, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Undecided